CLINICAL TRIAL: NCT02543723
Title: A Randomized Longitudinal Intervention Study to Assess the Efficacy and Feasibility of Telehealth-based Strategies to Increase Oral Chemotherapeutic Agent Medication Adherence and Health Literacy Among Cancer Patients.
Brief Title: Telehealth-based Strategies to Increase Oral Chemotherapeutic Agent Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Essie Torres, Assistant Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 53517
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Results first posted 2021-07-19 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Medication Adherence
Keywords: medication adherence, telehealth strategies, nurse coaching
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: We conducted a randomized control trial study of 150 subjects where subjects were randomly assigned to control or intervention arm. The Information-Motivation-Behavioral Skills Model of Adherence and the results of objective 1 guided this aim. Controls received the standard-of-care . The intervention arm received the standard-of-care and the nurse coach intervention. Specifically, we assessed whether a tailored nurse coaching intervention component will significantly improve medication adherence at higher rates as compared to the control group. The nurse coach intervention component involved individualized barriers/facilitators screening tool, educational tools, and regular contact with cancer patients via telephone calls across a six-month period.
Who Masked: Participant
Masking Description: Participants were randomized into the control or intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse Coach Intervention (Active Comparator): The nurse coach conducted an initial assessment with the participant and identified specific adherence strategies tailored to the participant's needs. The educational strategies include information about the patient's cancer treatment and expected outcomes; clear instructions about medication dosing schedule; what to do if a dose is missed or delayed; medication side effects and/or potential drug interactions; and review of cancer health literacy infographics. The behavioral skills and affective support strategies include coping strategies for side effects, skills for fitting medication regimen into daily routine, identifying a support network, communication skills for interacting with providers, and facilitating a positive perception for effective self-management experience. Patients received weekly phone calls from the nurse coach during the first month of the intervention, and then bi-monthly follow-up calls for the remainder of treatment or 6-month follow-up period.
  Interventions: Behavioral: Nurse Coach Intervention
- Control (No Intervention): Patients received standard of care.

INTERVENTIONS:
Behavioral: Nurse Coach Intervention — Participants randomized to the intervention 2 group a tailored nurse coach component. Participants will receive an initial session conducted by the nurse coach, via phone or in-person. Participants will receive weekly phone calls from the nurse coach during the first month of the intervention, and then bi-monthly follow-up calls for the remainder of treatment or 6-month follow-up period (whichever occurs first). The nurse coach will modify the intervention plan to address identified barriers to adherence at this time.
  Arms: Nurse Coach Intervention

SUMMARY:
Oral chemotherapeutic agents (OCAs) are increasingly being used as an alternative to traditional intravenous chemotherapy, and factors promoting this trend include increased survival times requiring long-term therapy, acceptability among patients, convenience, and cost savings due to reduced hospital time. Although OCAs are commonly preferred by patients, adherence to these medications vary. Suboptimal medication adherence leads to loss of treatment efficacy, increased toxicity, and increased health care costs. Thus, it is critical to develop and test interventions that effectively improve adherence to OCAs. Although the medication adherence literature has been criticized for methodological issues, some components of interventions have had promising results on adherence such as electronic monitored adherence feedback, cognitive-education, nurse-based interventions, and technology-based or telehealth strategies. The investigators propose to unify components of these effective approaches in a novel way to assess the efficacy and feasibility of two telehealth-based strategies (electronic medication-event monitoring with feedback and tailored nurse coaching which includes cognitive-education) in an effort increase OCA adherence among cancer patients who are at high-risk for non-adherence in rural eastern North Carolina.

DETAILED DESCRIPTION:
The purpose of this study is to improve cancer patient's adherence to their oral chemotherapy agents. We want to test whether a tailored nurse coaching intervention will significantly improve medication adherence as compared to a control group (standard-of-care). With strong support from our collaborators at the Vidant Cancer Care - Eddie and Jo Allison Smith Tower at Vidant Medical Center (VCC), study participants included cancer patients that were within their first two cycles of a new oral chemotherapy regimen at Vidant Medical Center/Leo W. Jenkins Cancer Center, which serves individuals throughout the 29 counties in rural eastern North Carolina (ENC).

Study Objectives:

Objective 1: To assess the barriers to, and facilitators of, adherence to oral chemotherapeutic agents among cancer patients who are at high-risk of non-adherence. Using the three-stage process of elicitation, intervention, and evaluation, we assessed factors that influenced non-adherence among this population. This formative qualitative assessment was accomplished by conducting interviews with English speaking cancer patients (N=25) and through key informant interviews/focus groups with cancer care providers (N=10). Objective 1 served as a baseline assessment to identify the unique factors that contribute to non-adherence and directly informed the development of tailored medication adherence strategies outlined in objective 2.

Objective 2. To test the effectiveness a telehealth adherence motivation strategy among cancer patients on oral chemotherapeutic agents who are at high-risk of non-adherence.

We conducted a randomized control trial study of 150 subjects where subjects were randomly assigned to control or intervention arm. The Information-Motivation-Behavioral Skills Model of Adherence and the results of objective 1 guided this aim. Controls received the standard-of-care. The intervention arm received the standard-of-care and the nurse coach intervention. Specifically, we assessed whether a tailored nurse coaching intervention component will significantly improve medication adherence at higher rates as compared to the control group. The nurse coach intervention component involved individualized barriers/facilitators screening tool, educational tools, and regular contact with cancer patients via telephone calls across a six-month period. We hypothesize that the nurse-coach intervention would be effective at increasing medication adherence. This hypothesis is supported by existing medication adherence literature that suggests a tailored intervention using multiple adherence strategies can potentially have a significant impact on increasing medication adherence.

ELIGIBILITY:
Inclusion Criteria:

1. New cycle or withing the first 3 cycles of OCAs
2. Ambulatory
3. Age 18 years or older
4. Able to consent for self
5. Able to read and speak English
6. Has a working cellphone or landline.

Exclusion Criteria:

1. Life expectancy <3 months as determined by oncologist
2. Current participation in a similar study or in investigational drug trials where adverse effects have not been fully elucidated
3. Presence of significant psychiatric or cognitive impairments as determined by oncologists and study teams.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-11-15 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Essie Torres, PhD, MPH, Principal Investigator — East Carolina University
Locations (1):
- Vidant Medical Center, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Patients received standard of care at this Regional Cancer Center.
Period: Overall Study
Arm/Group | Nurse Coach Intervention | Control
Started | 65 | 63
Completed | 65 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nurse Coach Intervention | Control | Total
Number analyzed (Participants) | 65 | 63 | 128
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 32 | 67
  >=65 years | 30 | 31 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (15.56) | 56 (48.08) | 53.25 (13.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 31 | 66
  Male | 30 | 32 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 30 | 63
  White | 29 | 33 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65 | 63 | 128
Cancer Health Literacy Test (CHLT-30) [Mean (Standard Deviation); unit: units on a scale] — The CHLT-30 measures cancer health literacy along a continuum with 0-30 representing the number of correct answers provided to the items. Continuous scores provided by the CHLT-30 do not allow to determine who has limited health literacy or put people in a category, but continuous scores indicate a degree of cancer health literacy, with the higher score indicating a higher degree of cancer health literacy.
  units on a scale | 20.17 (6.36) | 20.69 (6.15) | 20.42 (6.24)
Self-efficacy for Appropriate Medication Use Scale (SEAMS) [Mean (Standard Deviation); unit: units on a scale] — This is a validated 13-item self-report scale measuring patient confidence in the ability to take medications properly. This scale has 21 items scale, with scores ranging from 21-63, higher scores indicate higher level of self-efficacy for medication adherence.
  units on a scale | 58.16 (5.62) | 58.16 (6) | 58.16 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence at Baseline and 6-month Follow-up Period
Description: The participant's cancer medication adherence was taken at baseline and within a 6-month follow-up period. We measured the participant's self-efficacy with medication adherence increase with their OCAs using the SEAMS scale.
  SEAMS Scale: 21 items scale, ranges from 21-63, higher scores indicate higher level of self-efficacy for medication adherence.
Time Frame: Baseline and at 6 months
Population: Rural cancer patients taking oral cancer medications
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Nurse Coach Intervention; Control: Using the SEAMS to measure baseline and final (at 6 months)
Arm/Group | Nurse Coach Intervention | Control
Number analyzed (Participants) | 65 | 63
units on a scale | 59.4 (5.18) | 55.95 (9.34)

2. Secondary Outcome: Health Literacy at Baseline and 6-month Follow-up Period
Description: We measured the participant's cancer health literacy at baseline and at 6 months via the CHLT-30.
  The CHLT-30 measures cancer health literacy along a continuum with 0-30 representing the number of correct answers provided to the items. Continuous scores provided by the CHLT-30 do not allow to determine who has limited health literacy or put people in a category, with higher scores indicating a higher degree of cancer health literacy.
Time Frame: Baseline and at 6 months
Population: Rural cancer patients taking oral cancer medications
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Nurse Coach Intervention; Control: Using CHLT-30 to assess cancer health literacy in baseline and final (at 6 months)
Arm/Group | Nurse Coach Intervention | Control
Number analyzed (Participants) | 65 | 63
units on a scale | 22.95 (4.62) | 23.32 (8.36)

ADVERSE EVENTS:
Time Frame: 3 years (throughout the study)
Description: Our adverse events reporting description does not differ from the clinicaltrials.gov definition. We will be reporting All-Cause Mortality in this study.
Arm/Group | Nurse Coach Intervention | Control
All-Cause Mortality (participants affected / at risk) | 11/65 | 15/63
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/63
Other Adverse Events (participants affected / at risk) | 0/65 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT02543723/Prot_000.pdf